CLINICAL TRIAL: NCT05507853
Title: In the Joints or in the Brain? Exploring Central Sensitization in Pregnant Women and Its Role in Pain, Physical Activity, Functioning and Health Following Pregnancy
Brief Title: Exploring Central Sensitization in Pregnant Women
Status: Recruiting | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: VGFOUREG-939632
Record Dates: First submitted 2022-05-31; First posted 2022-08-19 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Pelvic Girdle Pain; Chronic Pain
MeSH Terms: conditions — Pelvic Girdle Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pelvic Girdle Pain (PGP) is reported by 50% of pregnant women and up to 11 years after pregnancy, 10% of women have persistent and per definition chronic PGP. Central (nervous system) sensitization that elicits pain hypersensitivity, may be one explanation.

The overall aim of this study is to explore features of central sensitization in pregnant women and its predictive ability on physical activity, functioning and health in women with PGP. Measurements of central sensitization will be done on two study groups, pregnant women with PGP and healthy controls. To identify women at risk to develop chronic pain in relation to a common pain experience ie PGP in pregnancy, may help us understand if central sensitization early in life explains why women develop chronic pain.

DETAILED DESCRIPTION:
Pelvic Girdle Pain (PGP) is reported by 50% (60000) of pregnant women yearly in Sweden. PGP is expected to disappear after delivery. However up to 11 years after pregnancy, 10% of women have persistent and per definition chronic PGP with large impact on their physical activity, functioning,and health. Central (nervous system) sensitization, defined as an amplification of neural signaling within the central nervous system that elicits pain hypersensitivity, may be one explanation why 10% of women develop postpartum chronic PGP and related physical inactivity.

The overall aim of this study is to explore features of central sensitization in pregnant women and its predictive ability on physical activity, functioning and health in women with PGP. Two study groups, pregnant women with PGP and healthy controls (including non-native Swedish) will be included through maternity care units and a blog. Measurements of primary outcome central sensitization will be done. To identify women at risk to develop chronic pain in relation to a common pain experience ie PGP in pregnancy, may help us understand if central sensitization early in life explains why women develop chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* pregnant (first time pregnant or previous experience of pregnancy)
* 18 years of age or older
* have a single foetus pregnancy
* be in gestational weeks 20-30
* able to read and understand Swedish or English

Exclusion Criteria:

* no history of a fracture or malignant disease in the back, pelvis, pelvic floor or hips
* no systemic disease of the musculoskeletal or the nervous system
* no diseases such as gestational diabetes or diabetes type 1 and 2, hypertension
* no obstetric complications
* no contradiction for tests.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant women at maternity care units and social media
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
central sensitization measured by Patient Pain Drawing | change from baseline (gestational week 20-30) at 6 weeks, at 6 months and at 12 months after delivery
  spreading of pain
central sensitization measured by conditioned pain modulation using an algometer and a occlusion cuff | change from baseline (gestational week 20-30) at 6 weeks, at 6 months and at 12 months after delivery
  Malfunctioning of descending nociceptive inhibitory pathways resulting in dysfunctional endogenous analgesia, assessed by a conditioned pain modulation (CPM)=
  1. PressurePainThresholds (PPT)is assed by a digital algometer at symtomatic (sacrum and lumbar paravertebral muscles and 2 remote locations)+at asymptomatic regions(web thumb-index, prox 1/3 calf )
  2. mechanism of CPM will be induced by inflating an occlusion cuff (conditioning stimulus) at the participant's left arm to a painful intensity. The occlusion cuff is inflated until 'the first sensation of pain' is reported. This cuff inflation is maintained for 30 sec. The participant is than asked to rate the pain intensity, as a result of cuff inflation at the left arm, on a NRS (0=no pain-10=worst pain). Next, the cuff inflation is increased or decreased until pain intensity at the left arm was rated as 3/10 on NRS. The PPT assessments are then repeated during maintenance of the cuff inflation and relaxation of the left arm.

SECONDARY OUTCOMES:
Pregnancy Physical Activity Questionnaire | change from baseline (gestational week 20-30) at 6 weeks, at 6 months and at 12 months after delivery
  Physical activity and exercise are measured by this self-administered questionnaire which provides assessment of four domains of physical activity; ''Sports and Exercises', ''Household and Caregiving'', 'Transportation''and ''Occupation'. Since it measures the frequency and the duration of the activities, (an intensity value assigned to each activity), the minimum values are 0 but here are no maximum values. The activities can be analyzed by type, by intensity or for the total energy expenditure.
Pelvic Girdle Questionnaire | change from baseline (gestational week 20-30) at 6 weeks, at 6 months and at 12 months after delivery
  Functioning. Minimum score 0 maximum score 100 where high scores mean worse outcome.
Patients Specific Functioning Scale | change from baseline (gestational week 20-30) at 6 weeks, at 6 months and at 12 months after delivery
  Two by the participant, self-chosen activities rated on a numeric rating scale. Minimum score 0 maximum score 10 where high scores mean better outcome
EuroQol 5-dimension questionnaire (EQ5D) | change from baseline (gestational week 20-30) at 6 weeks, at 6 months and at 12 months after delivery
  Health-related quality of life. Minimum score -0,59 and 1 maximum score where high scores mean better outcome
Work Ability Index | change from baseline (gestational week 20-30),at 12 months after delivery,
  Current work ability marked on a Numeric Rating Scale. Minimum score 0 maximum score 10 where high scores mean better outcome
Numeric Rating Scale for pain | change from baseline (gestational week 20-30) at 6 weeks, at 6 months and at 12 months after delivery
  pain intensity. Minimum score 0 maximum score 10 where high scores mean worse outcome
Numeric Rating Scale for concern | change from baseline (gestational week 20-30) at 6 weeks, at 6 months and at 12 months after delivery
  Concern. Minimum score 0 maximum score 10 where high scores mean worse outcome
Edinburgh Postnatal Depression Scale | change from baseline (gestational week 20-30) at 6 weeks, at 6 months and at 12 months after delivery
  Symptoms of depression. Minimum score 0 maximum score 30 where high scores mean worse outcome

OTHER OUTCOMES:
Fear-Avoidance Beliefs Questionnaire subscale on physical activity (FABQ-PA) | change from baseline (gestational week 20-30) at 6 weeks, at 6 months and at 12 months after delivery
  Fear avoidance beliefs about physical activity. Minimum score 0 maximum score 24 where high scores mean worse outcome
subscale Catastrophizing (CSQ-CAT),from the Coping Strategies Questionnaire | change from baseline (gestational week 20-30) at 6 weeks, at 6 months and at 12 months after delivery
  Catastrophizing thoughts. Minimum score 0 maximum score 52 where high scores mean worse outcome
General Self-Efficacy Scale | change from baseline (gestational week 20-30) at 6 weeks, at 6 months and at 12 months after delivery
  Self-efficacy. Minimum score 10 maximum score 40 where high scores mean better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Närhälsan Gibraltargatan, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided